CLINICAL TRIAL: NCT04597450
Title: Interventional, Randomized, Double-Blind, Crossover, Placebo-Controlled, Exploratory Study Investigating the Effects of Lu AG06466 on BOLD fMRI Signals and Sleep Parameters in Patients With PTSD
Brief Title: Lu AG06466 in Participants With Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 19364A
Record Dates: First submitted 2020-10-02; First posted 2020-10-22 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lu AG06466 (Experimental)
  Interventions: Drug: Lu AG06466
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AG06466 — Lu AG06466 - 30 mg/day, capsules, orally, once daily, one capsule will be taken daily for 15 days per treatment period
  Arms: Lu AG06466
Drug: Placebo — Placebo - capsules, orally, once daily, one capsule will be taken daily for 15 days per treatment period
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of Lu AG06466 after multiple doses of 30 milligrams (mg) in participants with PTSD.

DETAILED DESCRIPTION:
The crossover study consists of two treatment periods of 15 days duration. On Day -1 or Day 1 of Treatment Period 1, eligible participants will be randomized (1:1) to a sequence of treatments (either Lu AG06466-placebo or placebo-Lu AG06466) with 15 participants are planned per sequence. Each treatment period will be separated by a washout period of ≥7 and ≤14 days.

ELIGIBILITY:
Inclusion Criteria:

* The participant has PTSD, diagnosed according to Diagnostic and Statistical Manual Diploma in Social Medicine-5 (DSM-5), and confirmed by the Mini International Neuropsychiatric Interview (MINI).
* The participant has a Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) total score ≥28 at screening and baseline.
* The participant has alterations in arousal and reactivity, confirmed on CAPS-5.
* The participant has ongoing sleep disturbances, confirmed on CAPS-5.
* The participant is willing to discontinue all prohibited medications during the study and to complete a washout of psychotropic medication during the washout period.
* The participant does not have any magnetic resonance imaging (MRI) contraindications.

Exclusion Criteria:

* The index traumatic event that led to development of PTSD took place >15 years or <6 months before screening.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Functional Magnetic Resonance Imaging (fMRI) Data: Mean Blood Oxygen Level Dependent (BOLD) Percent Signal Change During Facial Affect Recognition Task | Day 15
  fMRI parameter estimates (β-contrasts) will be extracted per participant/treatment period from task-related regions of interest (ROIs) under task-specific contrast, Facial Affect Recognition Task
Functional Magnetic Resonance Imaging (fMRI) Data: Mean Blood Oxygen Level Dependent (BOLD) Percent Signal Change During Threat Processing Task | Day 15
  fMRI parameter estimates (β-contrasts) will be extracted per participant/treatment period from task-related regions of interest (ROIs) under task-specific contrast, Threat Processing Task
Functional Magnetic Resonance Imaging (fMRI) Data: Mean Blood Oxygen Level Dependent (BOLD) Percent Signal Change During Card Guessing Task | Day 15
  fMRI parameter estimates (β-contrasts) will be extracted per participant/treatment period from task-related regions of interest (ROIs) under task-specific contrast, Card Guessing Task
Skin Conductance Response (SCR) During fMRI Tasks | Day 15
  SCR in micro-Siemens
Skin Conductance Response (SCR) During the Threat Processing Task | Day 14
  SCR in micro-Siemens
Behavioural Measures During fMRI Tasks | Day 15
  Behavioural Response: behavioural measures rated on a 3-point scale
Behavioural Measures During the Threat Processing Task | Day 14
  Behavioural Response: behavioural measures rated on a 3-point scale
Sleep, Polysomnography (PSG) Parameters: Total Sleep Time (TST) | Day 12-13
  TST in minutes
Sleep, Polysomnography (PSG) Parameters: Sleep Efficiency (SE) | Day 12-13
  SE in percent
Sleep, Polysomnography (PSG) Parameters: Wake-Time After Sleep-Onset (WASO) | Day 12-13
  WASO in minutes
Sleep, Polysomnography (PSG) Parameters: Sleep Onset Latency (SOL) | Day 12-13
  SOL in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Collaborative NeuroScience Network LLC, Long Beach, California, United States